CLINICAL TRIAL: NCT04002726
Title: Developing and Evaluating Trachoma Diagnosis Training Tools in Preparation for the Trachoma Elimination Endgame: Investigating the Effectiveness, Acceptability and Feasibility of an App-based Versus Slide-based IGA Test for Trachoma Graders
Brief Title: App-based Versus Slide-based Inter-grader Agreement (IGA) Test for Trachoma Graders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); Federal Minstry of Health of Ethiopia (Other Government); Jos University Teaching Hospital (Other); University College London Hospitals (Other); RTI International (Other); Sightsavers (Unknown); World Health Organization (Other); Pan American Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2019-KEP-284 - 1
Record Dates: First submitted 2019-06-19; First posted 2019-07-01 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-05

CONDITIONS: Trachoma
MeSH Terms: conditions — Trachoma | interventions — Immunoglobulin A; Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group Aa (Active Comparator): Allocated to do the app-based training. Allocated to do the app-based classroom IGA test first, and the slide-based test second.
  Interventions: Other: Inter-grader agreement (IGA) app
- Group As (Active Comparator): Allocated to do the app-based training. Allocated to do the slide-based classroom IGA test first, and the app-based test second.
  Interventions: Other: Inter-grader agreement (IGA) app
- Group Sa (Active Comparator): Allocated to do the slide-based training. Allocated to do the app-based classroom IGA test first, and the slide-based test second.
  Interventions: Other: Inter-grader agreement (IGA) app
- Group Ss (Active Comparator): Allocated to do the app-based training. Allocated to do the slide-based classroom IGA test first, and the app-based test second.
  Interventions: Other: Inter-grader agreement (IGA) app

INTERVENTIONS:
Other: Inter-grader agreement (IGA) app — A smartphone-based app with images of conjunctivae for trachoma grading training purposes.

SUMMARY:
Trachomatous inflammation-follicular (TF) is diagnosed by looking for clinical signs of infection of everted eyelids (conjunctivae) of children.

The overall objective of this project is to investigate the effectiveness, acceptability and feasibility of an app-based versus slide-based IGA for trachoma graders.

Fieldwork will take place during routine Tropical Data trainings. A non-inferiority randomised controlled trial design will be employed, with grader trainees randomised to app- or slide-based training, and then to app- or slide-based IGA testing. The training and IGA testing method will be compared with field IGA test score to determine which method best predicts passing the field IGA test.

DETAILED DESCRIPTION:
Trachoma graders are currently trained using either slide- or app-based testing systems. The investigators want to formally assess whether the app-based training and testing system leads to better field-based diagnosis than the slide-based training and testing system. The investigators will also ask participants for their views on acceptability of the two systems and conduct a cost-consequences analysis of the two systems.

Objectives and approach:

1.1 To compare the two classroom IGA tests (app-based and slides-based) in terms of their ability to predict trainee success in the field IGA test.

1.2 To assess whether the kappa score threshold for the classroom IGA tests is appropriate.

1.3 To conduct a cost-consequences analysis of the training systems in order to effectively target the use of an app-based assessment and training system.

1.4 To investigate whether grader trainee characteristics have an impact on trainee performance in the IGA tests.

1.5 To obtain feedback on the app-based system's usability and acceptability. 1.6 To compare the two classroom IGA training methods (app-based and slides-based) in terms of classroom IGA test (app-based and slides-based) outcome and field IGA test outcome.

ELIGIBILITY:
Inclusion Criteria:

* All trainers and trainee graders who attend selected Tropical Data training events will be eligible for inclusion in the study.

Exclusion Criteria:

* Individuals who do not provide consent are not eligible for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Classroom IGA success | 1 day
  The proportion of participants successfully passing (kappa ≥0.7) the app-based IGA.
Classroom IGA success | 1 day
  The proportion of participants successfully passing (kappa ≥0.7) the slide-based IGA.
Field IGA success | 3 days
  The correlation between classroom IGA score and field IGA score
Field IGA success | 3 days
  The proportion of participants who successfully pass the classroom IGA test (kappa ≥0.7) who also successfully pass the field-based IGA test (kappa ≥0.7)

SECONDARY OUTCOMES:
Trainee characteristics | 5 days
  Association (reported as proportions, unadjusted and adjusted odds ratios) between trainee characteristics and the probability of successfully passing classroom IGA test
Trainee characteristics | 5 days
  Association (reported as proportions, unadjusted and adjusted odds ratios) between trainee characteristics and the probability of successfully passing the field IGA test
Acceptability and feasibility (common themes from focus group discussions) of app versus slide-based training. | 45 minutes
  Common themes, as determined through thematic analysis of focus group discussion transcripts, relating to acceptability and feasibility of app versus slide-based training.
Acceptability and feasibility (common themes from focus group discussions) of app versus slide-based IGA testing. | 45 minutes
  Common themes, as determined through thematic analysis of focus group discussion transcripts, relating to acceptability and feasibility of app versus slide-based IGA testing.
Cost of app versus slide-based training | 5 days
  Cost (overall and broken down by category: personnel; supplies; transit; telecommunications) of app versus slide-based training
Cost of app versus slide-based IGA testing | 5 days
  Cost (overall and broken down by category: personnel; supplies; transit; telecommunications) of app versus slide-based IGA testing

CONTACTS AND LOCATIONS:
Overall Officials: Emma Harding-Esch, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Arusha region, Arusha, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared with relevant study team members for the purposes of data analysis. Data Transfer Agreements will be completed, where appropriate.
Supporting Information: Study Protocol
Time Frame: Data will be shared with team members as they are collected.
Access Criteria: Data access requests from outside the study team for the specified data analyses will be reviewed by the Principal Investigator. Requestors will be required to sign a Data Access Agreement.